CLINICAL TRIAL: NCT06364267
Title: Randomized Double Blind Phase II Trial of Baby Exemestane vs Baby Tamoxifen in Post-menopausal Women at High Risk for Breast Cancer.
Brief Title: Low Dose Exemestane vs Low Dose Tamoxifen in Post-menopausal Women at High Risk for Breast Cancer.
Acronym: BabyTears
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea DeCensi (Other)
Collaborators: Dana-Farber/Brigham and Women's Cancer Center (Other); Herbert Irving Comprehensive Cancer Center (Other); Istituto Europeo di Oncologia (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Andrea DeCensi, Director of Medicin Department and Oncology Division, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BabyTears; 2024-520004-26-00 (EU CTIS Number)
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer, menopause, exemestane, tamoxifen, MenQol, Low dose; babytam, babyexe
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM 1 (Experimental): BabyEXE Arm, 25 mg eod, typically every odd day of the monthly calendar for 12 months.
  Interventions: Drug: Exemestane 25 MG
- ARM 2 (Experimental): BabyTAM Arm, 10 mg eod, typically every odd day of the monthly calendar for 12 months
  Interventions: Drug: Tamoxifen 10 MG

INTERVENTIONS:
Drug: Tamoxifen 10 MG — Blinded tamoxifen 10 mg every other day
  Arms: ARM 2
Drug: Exemestane 25 MG — Blinded exemestane 25 mg every other day
  Arms: ARM 1

SUMMARY:
The purpose of the study is to to compare low dose of exemestane (babyexe) versus low dose of tamoxifen (babytam) in terms of change of quality of life from baseline to 12 months.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind phase II trial.

Eligible patients will be randomized in a 1:1 ratio to:

ARM 1: BabyEXE Arm, 25 mg eod, typically every odd day of the monthly calendar for 12 monthsor unless progression, SAE, medical decision, patient withdrawal occur.

ARM 2: BabyTAM Arm, 10 mg eod, typically every odd day of the monthly calendar for 12 months or unless progression, SAE, medical decision, patient withdrawal occur.

Blinding will be guaranteed by over-encapsulation of active tablet agents with an AA capsule in a 6-month bottle.

In both arms, treatment should begin within 30 days from randomization. Exemstane and Tamoxifen will be provided for free by the Study Sponsor.

After study completion, participants will be unblinded and treated according to local guidelines. Clinical visit will be performed every 6 months (±14 days) with physical examination vital signs and weight and girth measurement, ECOG PS, MENQOL questionnaire (0, 6, 12 months), review of self-reported compliance, concomitant medications, AEs assessment, and physical exam. Telephone/video contact may be allowed at 3 and 9 months, whereas baseline, 6 months and 12 months visits are necessary for blood collection and biomarker assessment. Blood serum for centralized storage at IEO, Milan, Italy, will be collected at different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post- menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   Any of the following criteria must be met:
   1. Recent (within 12 months from date of consent form signature) histologic diagnosis of ER+ve (>5%) DCIS (patients with DCIS should have undergone breast-conserving therapy i.e. lumpectomy to remove the tumor with negative surgical margins followed by radiotherapy) or diagnosis within 3 years of HRL (ADH, LCIS, ALH), or:
   2. At least 3% breast cancer risk at 5 years (or 5% risk at 10yrs) per one of the following risk models: the Breast Cancer Surveillance Consortium risk calculator V3 or Tyrer-Cuzick model V8 or:
   3. Known carriers of a germline pathogenic/likely pathogenetic variant in the following moderate penetrance genes (CHEK2 or ATM), or women with chest wall irradiation before age of 30 years.
2. Eastern Cooperative Oncology Group - Performance Status (ECOG-PS) 0-1.
3. Able to swallow oral medications.
4. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Specifically, all cancers diagnosed since 3 years or longer except for breast and endometrial are eligible.
5. Ability to understand and the willingness to sign a written informed consent document.
6. Mammography performed up to 6 months before the trial consent form signature.
7. DEXA performed up to 12 months before the trial consent form signature.
8. Patients with life expectancy ≥ 10 years.
9. Patients with normal liver function tests and blood cell count.
10. Negative gynaecological examination performed up to 6 months before the trial consent form signature.

Exclusion Criteria:

1. Pre/perimenopausal women
2. History of DVT or PE.
3. Endometrial cancer.
4. Macular disorders.
5. Inability to comply with study procedures.
6. Prior use of antiestrogens within 12 months from the date of the trial consent form signature.
7. Use of hormone replacement therapy (HRT) within 3 months from the date of the trial consent form signature.
8. Severe osteoporosis (T score ≤ 2.5 at either spine or hip), or recent vertebral fracture (within 6 months) not treated with zolendronic acid or denosumab.
9. Use of terbinafine, quinidine, cinacalcet, rifampicin, phenytonin, carbamazepine, phenobarbital, and St. John's wort, warfarin, erythromycin, cyclosporin, nifepidine and any concomitant coumarin-type anticoagulant therapy.
10. Patients with moderate or severe renal impairment.
11. Patients with a known hypersensitivity to study drugs.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life MEnQol | 12 months
  The primary endpoint is the difference between arms in the score of overall domain of MENQOL after 12 months of treatment.

SECONDARY OUTCOMES:
Sex hormones | 12 months
  The difference in sex hormones (free estradiol: estradiol/SHBG) and IGF system (IGF-I, IGFBP-3 and their ratio) after 12 months, as surrogate endpoint biomarkers.
MenQol score domain | 6 months
  The difference between arms in the overall MENQOL score domain after 6 months of treatment.
Sex hormones | 6 months
  The difference in sex hormones (free estradiol: estradiol/SHBG) and IGF system (IGF-I, IGFBP-3 and their ratio) after 6 months, as surrogate endpoint biomarkers.
Other domains of MenQol | 6 and 12 months
  The difference between arms individual domains of MENQOL (physical, sexual, psychosocial, vasomotor) at 6 and 12 months
Safety profile | 6 and 12 months
  The difference between arms of safety profile according to CTCAE v.5 at 6 and 12 months.
PMAS | 6 and 12 months
  The difference between arms at 6 and 12 months in PMAS, Promise Medication Adherence Scale, a validated tool to measure pill adherence.
BPI | 6 and 12 months
  The difference between arms on BPI Brief Pain Inventory at 6 and 12 months.
Bone biomarker | 6 and 12 months
  The difference between arms in C-telopetide at 6 and 12 months
Customer satisfatcion | Screening
  Patient uptake at screening/baseline phase will be measured with a questionnaire including factors related to breast cancer worry and presence of life style risk factors, and participant satisfaction for study explanation.
Exemestane toxicity | 12 months
  Toxicity of babyexe in comparison with full dose historical controls treated in the adjuvant setting will also be evaluated

OTHER OUTCOMES:
MMG risk score | 12 months
  Change at 12 months of risk score using an image derived artificial intelligence risk model for digital mammography.
MMG density | 12 months
  Change at 12 months of mammographic density using an image derived artificial intelligence model.
HOMA | 6 and 12 months
  Change at 6 and 12 months of HOMA index
Hs-CRP | 6 and 12 months
  Change at 6 and 12 months of hs-CRP
Adipokines | 6 and 12 months
  Change at 6 and 12 months of adipokines (adiponectin and leptin).
Bone density | 12 months
  Difference between arms in the change in T-score of lumbar spine and femur as measured by DEXA at 12 months.
BMI | 6 and 12 months
  Difference between arms at 6 and 12 months in the changes in primary and secondary endpoints by BMI in kg/m^2
Other biomarkers | 6 and 12 months
  Menopausal symptoms and biomarker levels by serum drug and metabolite levels at 6 and 12 months in each arm. Tamoxifen, 4-OH-tamoxifen, endoxifen, other tamoxifen metabolites, exemestane and 17OH-exemestane will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea U De Censi, MD, Study Chair — Ente Ospedaliero Ospedali Galliera
Locations (1):
- E.O. Ospedali Galliera, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: No